CLINICAL TRIAL: NCT06828783
Title: Development of Anti-Ageing Health Supplement From Subcritical Water Extraction of Zingiber Officinale Roscoe (Ginger) Bioactive Compounds
Brief Title: Anti-Ageing Health Supplement From Ginger Extracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UKM PPI/111/8-JEP-2022-395
Record Dates: First submitted 2025-02-05; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Ageing Signs; Cognitive Decline; Musculoskeletal
MeSH Terms: conditions — Cognitive Dysfunction | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented (Experimental): Each participant will be supplemented with ginger-based capsules.
  Interventions: Dietary Supplement: ginger extract
- Placebo (Placebo Comparator): Each participant will be supplemented with placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: ginger extract — Participants will receive a ginger-based capsule
  Arms: Supplemented
Other: Placebo — Participants will receive a placebo capsule
  Arms: Placebo

SUMMARY:
This study examines the development and efficacy of a health supplement derived from ginger using water extraction. Designed to address aging-related issues such as muscle loss (sarcopenia) and cognitive decline, the capsule's safety and effectiveness were evaluated through clinical trials. Stability testing ensured the capsules maintained their quality under various environmental conditions. Clinical trials further assessed the supplement's antioxidant and anti-inflammatory properties. The findings support its potential benefits for elderly health and aging-related challenges.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male
* Blood chemistry results specifically Blood Urea Nitrogen (BUN), Serum Creatinine, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-glutamyl transpeptidase (GGTP), Total Bilirubin and alkaline phosphatase and urinalysis results, specifically urine pH, protein, glucose, ketone, and bilirubin levels within +/- 20% of normal value indicated in the lab report.
* Individuals are willing to maintain their exercise habits and dietary patterns throughout the trial
* No allergy to ginger
* Provide written informed consent before screening
* Subject is willing and able to comply with the study visit schedule and procedure, geographic proximity (investigator's discretion) that allows adequate follow-up
* Subjects understand the study protocol and sign informed consent forms

Exclusion Criteria:

* Use of dietary supplements within one week of Day 0. Supplements include any ginger (Zingiber officinale, ginger root, black ginger, zingiberis rhizoma) vitamins, minerals, and herbal products, including herbal drinks.
* Presence of, or clinically significant history of, cancer, cardiovascular, endocrine, kidney, liver, lung, gastrointestinal, metabolic disorder, absorption disorder such as Celiac or Crohn's disease and/or any other chronic health condition such as diabetes identified from the findings of the interview.
* Presence of gallstones or history of gallbladder disease.
* Presence or history of diabetes.
* Presence of cardiovascular disease and hypertension with inconsistent medication regimen, unstable conditions, and without proper physician's - Ten hours before the blood and urine sample collection, subjects should refrain from using medications such as statins (e.g., simvastatin, fluvastatin), NSAIDS including paracetamol, aspirin, nitric oxide (eNOS) activators or inhibitors (e.g., selegiline, Viagra), and angiotensin II receptor blocker (e.g., Telmisartan (blood pressure)) or take any of these medications
* Subjects with vegan diet
* Current smoker or used to smoke in the past 3 months
* Subject for surgery or had undergone surgery in the past 3 months History of bleeding tendencies or any condition predisposing to bleeding e.g. thrombocytopenia, abnormal liver function, liver disease (e.g. chronic hepatitis), gastrointestinal ulcers
* Subjects who have significantly changed their physical activity in the past 2-4 weeks or who intend to change them during the study
* Participation in another clinical trial within 30 days of enrolment into the study.
* History or current abuse of nicotine, drugs, or alcohol, or intake > 3 alcoholic beverages per day

Ages: 48 Years to 63 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants are often preferred in clinical trials due to their more stable physiology, reducing variability in results. Hormonal fluctuations in females from menstrual cycles, pregnancy, and menopause can affect metabolism, drug absorption, and inflammatory responses, complicating data analysis. Men also have higher muscle mass and lower fat percentage, influencing the effects of drugs or supplements on muscle strength and metabolism. Additionally, avoiding potential hormonal interactions and reproductive health risks makes early-phase trials safer and more controlled. While modern trials aim for gender balance, male participants help minimize biological variability and ensure clearer outcomes.
Enrollment: 90 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle mass | Baseline and 24 weeks after supplementation
  Appendicular lean mass in kilograms, kg will be measured using Dual-Energy X-ray Absorptiometry, (DEXA)
Fat mass | Baseline and 24 weeks after supplementation
  Fat mass in gram, g will be measured using Dual-Energy X-ray Absorptiometry, (DEXA)
Bone mineral content (BMC) | Baseline and 24 weeks after supplementation
  Bone mineral content in gram, g will be measured using Dual-Energy X-ray Absorptiometry, (DEXA)
Gait speed test | Baseline and 24 weeks after supplementation
  Gait speed will be measured in meters per second (m/s). Participants will complete three walking trials, with each trial timed over a 6-meter distance to record gait speed in seconds.
Handgrip strength | Baseline and 24 weeks after supplementation
  Evaluation of hand grip strength will be conducted using a dynamometer. Participants will be instructed to grip the dynamometer. The values will be recorded in kilograms (kg)
Cognitive function | Baseline and 24 weeks after supplementation
  The assessment instrument, the Montreal Cognitive Assessment (MoCA) test will be administered. The evaluation involves assessing participants through questions and instructions covering executive and spatial cognitive domains. The maximum score is 30. A score of 26 and above indicates no cognitive impairment.
Recall memory function | Baseline and 24 weeks after supplementation
  The Rey Auditory Verbal Learning Test (RAVLT) will be utilized. The RAVLT includes two distinct word lists (A and B). Participants will recall the items from list A over five trials (Memory A1 to A5). Following this, an interference list (list B), comprising 15 unrelated nouns, will be introduced, and participants will attempt to recall as many words as possible from it. Subsequently, participants will be asked to recall the words from list A (Delayed recall/Memory A6) without the examiner repeating the list. The number of correctly recalled words for each trial will be totaled to generate a score.
  Total Learning Score (Sum of Trials A1-A5) to indicate normal performance: 45-65, Mild Cognitive Impairment: 30-45, dementia: below 30. For delayed recall score (M6), to indicate normal performance: ≥8-12 words recalled, Mild Cognitive Impairment: 4-7 words recalled, and dementia: ≤3 words recalled.
Working memory function | Baseline and 24 weeks after supplementation
  The Digit Span Test involves recalling numbers in the same order (forward), reverse order (backward), or ascending order (sequencing). The test starts with short sequences and increases in length to assess memory capacity. A higher score (20 - 30) indicates better cognitive function, while a lower score (0 - 19) may suggest attention or memory issues. The total score is 30.

SECONDARY OUTCOMES:
Blood pressure | Baseline and 24 weeks after supplementation
  Blood pressure in mmHg using Sphygmomanometer
C-Reactive protein (CRP) | Baseline and 24 weeks after supplementation
  CRP level in serum will be measured using Particle-Enhanced Turbidimetric Immunoassay (PETIA) in mg/dL
Untargeted metabolomics for metabolite identification | Baseline and 24 weeks after supplementation
  Untargeted metabolomics for metabolite identification will be conducted using a Quadrupole-Orbitrap Mass Spectrometer. It begins with sample preparation, followed by liquid chromatography (LC) to separate metabolites before mass spectrometry analysis. Data is then processed using MetaboAnalyst to extract, align, and annotate metabolites by matching them to the Human Metabolome Database (HMDB) and Kyoto Encyclopedia of Genes and Genomes (KEGG) databases. The Principal Component Analysis (PCA) will be applied to identify significant metabolites, which are subsequently mapped to biological pathways for interpretation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz, UKM Medical Centre, Cheras, WP Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication and ending 3 years after the publication of results
Access Criteria: The Principal Investigator will review the request.